CLINICAL TRIAL: NCT06414525
Title: Effect of Abdominal Massage Versus Visceral Manipulation on Constipation Status and Quality of Life in Adults
Brief Title: Effect of Abdominal Massage Versus Visceral Manipulation on Constipation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mennat Allah Mohamed Ali Ahmed, head of department of physical therapy AboKhalefa hospital, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: constipation
Record Dates: First submitted 2024-05-06; First posted 2024-05-16 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Constipation Chronic Idiopathic
Keywords: chronic idiopathic constipation; abdominal massage; visceral manipulation; quality of life
MeSH Terms: interventions — Diet; Bathroom Equipment

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Abdominal massage (Active Comparator): The technique involves stroking and kneading the abdomen in a consistent pattern.
  Interventions: Other: abdominal massage
- visceral manipulation (Active Comparator): The technique involves visceral connective tissue manipulation.
  Interventions: Other: visceral manipulation
- control (Active Comparator): instructions on daily, dietary, toilet, and physical activity habits
  Interventions: Other: instructions on daily, dietary , toilet , and physical activity habits

INTERVENTIONS:
Other: abdominal massage — It will include patients that will receive abdominal massage; the frequency and duration of the massage will be arranged as 3 sessions per week, with each session lasting an average of 20-25 minutes for 6 weeks.
  Arms: Abdominal massage
Other: visceral manipulation — It will include patients that will receive visceral manipulation; the frequency and duration of the technique will be arranged as 3 sessions per week, with each session lasting an average of 20-25 minutes for 6 weeks.
  Arms: visceral manipulation
Other: instructions on daily, dietary , toilet , and physical activity habits — It will include patients that will receive behavioral therapy: defecation mechanism and informing about negative attitudes and behaviors towards defecation), lifestyle advice (diet, water consumption, fiber food, etc.), teaching effective defecation posture, and timed toilet training.
  Arms: control

SUMMARY:
The study compares the effect of abdominal massage vs. visceral manipulation on constipation status and quality of life in adults.

Chronic idiopathic constipation (CIC) is considered a common functional bowel disorder characterized by difficult, infrequent, and/or incomplete defecation. It has a great impact on the quality of life and on the healthcare system and represents an important financial strain .

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sex with age ranges (20-40) years old.
* having a diagnosis of functional constipation according to Rome IV criteria onset of constipation symptoms from 6-12 months .
* having body mass index 18.5-29.9 kg/m2 , waist height ratio </=0.5
* Subjects bothered by their constipation

Exclusion Criteria:

* Pregnancy.
* Having comorbidities (chronic pelvic pain, neurological (Parkinson's, multiple sclerosis, spinal cord lesion, etc.), metabolic / endocrine (diabetes mellitus, hypercalcemia, hypothyroid, etc.), cardiorespiratory diseases
* Health problems which may prevent standing from sitting, walking (orthopedic, neurological, cardiorespiratory, etc.)
* Malignancy, acute inflammation, intestinal tumor
* History of gastrointestinal and pelvic surgery or spinal surgery other than cholecystectomy, appendectomy, or hysterectomy
* Visual, auditory or cognitive problems which may prevent participation to the study.
* Tumor, presence of skin problems in the application area
* Presence of laxative use for functional constipation in the last four weeks or patients on laxative therapy.
* Alarm symptoms (unexplained, more than 10% weight loss in 3 months, hemorrhoids and anal fissures, rectal bleeding, family history of colon cancer)

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Constipation Severity Instrument (CSI) | 6 weeks
  Constipation Severity Instrument (CSI) will be used to evaluate the severity of the constipation. The Constipation Severity Instrument is a 16-item patient-reported outcome measure that investigates symptoms of constipation based on frequency, severity, and bother of symptoms. CSI consists of three subscales: obstructive defecation, colonic inertia, and pain.
  Higher scores of CSI indicate more severe constipation.
Constipation Assessment Scale | 6 weeks
  Constipation assessment scale will be used to evaluate the severity of the constipation. The constipation assessment scale is a eight-item scale that assess the presence and severity of constipation.
  The patient rates each constipation item on a three-point scale (no problem to severe problem). Total scores range from 0 (no constipation) to 16 (worst possible constipation).
Patient Assessment of Constipation- Quality of Life (PAC-QOL) Questionnaire | 6 weeks
  Patient Assessment of Constipation Quality of Life Questionnaire (PAC-QOL) will be used to evaluate quality of life. PAC-QOL consists a total of 28 items in four subscales: worries and concerns (11 items), physical discomfort (4 items), psychosocial discomfort (8 items), and satisfaction (5 items). Higher scores of PAC-QOL indicate more negative effects of constipation on the quality of life.
Bowel Function Index | 6 weeks
  (Scale 0 - 100), will be calculated as the mean of three variables (ease of defecation, feeling of incomplete bowel evacuation, and personal judgement of constipation) was developed to evaluate bowel function.

CONTACTS AND LOCATIONS:
Locations (1):
- Abo Khalefa emergency hospital, Ismailia, Egypt